CLINICAL TRIAL: NCT06182020
Title: The Effect of Integrated Care Involving Peripheral Functional Magnetic Stimulation and Nutritional Supplement for Age-related Sarcopenia
Brief Title: Effect of Integrated Care Involving Peripheral Functional Magnetic Stimulation for Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202309121RIND
Record Dates: First submitted 2023-11-23; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Functional magnetic stimulation
MeSH Terms: conditions — Sarcopenia | interventions — Dietary Supplements; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated care (Experimental): Participants in this group will receive both the peripheral functional magnetic stimulation to both the upper and lower limbs and nutritional supplement for consecutive 8 weeks.
  Interventions: Device: Peripheral functional magnetic stimulation (ISKRA MEDICAL TESLA Former prestige Magneto therapy); Dietary Supplement: Nutritional supplementation (ENSURE HIGH CALCIUM)
- Usual care (Active Comparator): Participants in this group will receive an educational DVD and one session of oral instructions on general care and exercise suggestions for sarcopenia.
  Interventions: Behavioral: Education

INTERVENTIONS:
Device: Peripheral functional magnetic stimulation (ISKRA MEDICAL TESLA Former prestige Magneto therapy) — The peripheral functional magnetic stimulation will be conducted 30 minutes a session, 2 sessions per week, for consecutive 8 weeks. The stimulation will be placed over bilateral forearm flexor muscles and bilateral thighs over rectus femoris muscles.
  Arms: Integrated care
Dietary Supplement: Nutritional supplementation (ENSURE HIGH CALCIUM) — The nutritional supplementation includes 7 cans of "ENSURE HIGH CALCIUM" per week for 8 consecutive weeks.
  Arms: Integrated care
Behavioral: Education — The education includes a DVD and one session of oral instructions on general care and exercise suggestions for sarcopenia.
  Arms: Usual care

SUMMARY:
The goal of this clinical randomized trial is to test whether an integrated care involving peripheral functional magnetic stimulation and nutritional supplement is beneficial in population with age-related sarcopenia, as compared to usual care.

DETAILED DESCRIPTION:
We will recruit participants with sarcopenia or possible sarcopenia. The participants will be divided into 2 groups. One group, the "integrated care" group, will receive both the peripheral functional magnetic stimulation to both the upper and lower limbs and nutritional supplement for consecutive 8 weeks. The other group, the "usual care" group, will receive an educational digital versatile disc (DVD) and a handbook for exercise suggestions on sarcopenia. We will compare before and after the intervention about the body composition, handgrip strength, 5-time chair stand test, 6-meter walk, and blood test for C-reactive protein and other cytokines related to sarcopenia. The participant's nutritional condition, activity level, life quality will also be analyzed via questionnaires before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age from 65 to 90
* Can walk independently for over 15 minutes
* Diagnosed with possible sarcopenia or sarcopenia (by Asian Working Group for Sarcopenia: 2019 Consensus Update onSarcopenia Diagnosis and Treatment)

Exclusion Criteria:

* Cognitive impairment
* History of cerebrovascular disease
* Deep vein thrombosis
* Malignancy under treatment
* Coagulopathy
* Serious orthopedic condition over limbs
* Inability to walk independently without assistive device
* Any other conditions not suggested to performance exercise
* Medical implants (e.g. pacemaker, defibrillator, deep brain nerve stimulation, infusion pump, etc.)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Body composition | Before the intervention, and 1-2 weeks after the 8-week intervention
  We use dual energy x-ray absorptiometry to evaluate the muscle mass (kg/m2) in the subjects.
Handgrip strength | Before the intervention, and 1-2 weeks after the 8-week intervention
  We use a dynamometer to measure the handgrip strength (kg)
5-time chair stand test | Before the intervention, and 1-2 weeks after the 8-week intervention
  We measure the time of a subject to transfer from a seated to a standing position and back to sitting five times.
6-meter walk | Before the intervention, and 1-2 weeks after the 8-week intervention
  We measure the time of a subject to walk with the usual speed straightly for 6 meters.

SECONDARY OUTCOMES:
Leg circumference | Before the intervention, and 1-2 weeks after the 8-week intervention
  We measure the largest calf circumference with seated position with knee flexed in 90 degrees.
Cytokines related to sarcopenia | Before the intervention, and 1-2 weeks after the 8-week intervention
  We will check the concentrations of cytokines including the c-reactive protein from our subjects.
Nutritional status | Before the intervention, and 1-2 weeks after the 8-week intervention
  We use the questionnaire Mini Nutritional Assessment to evaluate the subjects' nutritional status.
Activity level | Before the intervention, and 1-2 weeks after the 8-week intervention
  We use the International Physical Activity Questionnaire to evaluate the subjects' activity levels.
Life quality | Before the intervention, and 1-2 weeks after the 8-week intervention
  We use the EuroQol-5 dimensions (EQ-5D) and Taiwan Short Form-36 questionnaires to evaluate the subjects' health life quality.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yu Chi, Principal Investigator — National Taiwan University Hospital Bei-Hu Branch
Locations (1):
- National Taiwan University Hospital Bei-Hu Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No